CLINICAL TRIAL: NCT07230639
Title: Node-Sparing Hypofractionated Radiotherapy Plus Chemotherapy and PD-1 Inhibitor in pMMR/MSS High-Risk Locally Advanced Colon Cancer: A Prospective, Randomized, Phase II Trial
Acronym: MODIFI-CC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, MD PHD, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC502
Record Dates: First submitted 2025-09-16; First posted 2025-11-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Neoadjuvant Therapies; Immune Checkpoint Therapy; Radiotherapy
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25Gy/5F Radiotherapy Group (Experimental): Node-Sparing Short-Course RT (25Gy/5F) followed by sequential Chemotherapy and PD-1 inhibitor as total neoadjuvant therapy.
  Interventions: Combination Product: Node-Sparing Radiotherapy(25Gy/5F) plus Chemotherapy and PD-1 inhibitor
- 24Gy/4F Radiotherapy Group (Experimental): Node-Sparing Short-Course RT (24Gy/4F) followed by sequential Chemotherapy and PD-1 inhibitor as total neoadjuvant therapy.
  Interventions: Combination Product: Node-Sparing Radiotherapy(24Gy/4F) plus Chemotherapy and PD-1 inhibitor

INTERVENTIONS:
Combination Product: Node-Sparing Radiotherapy(25Gy/5F) plus Chemotherapy and PD-1 inhibitor — Patients will receive node-sparing modified short-course radiotherapy(25Gy/5F), followed by 4 cycles of CAPOX chemotherapy combined with a PD-1 inhibitor. After neoadjuvant treatment, patients will undergo surgery.
  Arms: 25Gy/5F Radiotherapy Group
Combination Product: Node-Sparing Radiotherapy(24Gy/4F) plus Chemotherapy and PD-1 inhibitor — Patients will receive node-sparing modified short-course radiotherapy(24Gy/4F), followed by 4 cycles of CAPOX chemotherapy combined with a PD-1 inhibitor. After neoadjuvant treatment, patients will undergo surgery.
  Arms: 24Gy/4F Radiotherapy Group

SUMMARY:
Most colorectal cancers are microsatellite stable (MSS) or mismatch repair-proficient (pMMR) subtypes, which show limited efficacy to PD-1 inhibitors. Radiotherapy can enhance the release of tumor-associated antigens, thereby improving the responsiveness of pMMR/MSS colorectal cancers to PD-1 blockade. Tumor-draining lymph nodes (TDLNs) are critical sites where PD-1 inhibitors exert their antitumor effects; however, previous studies have reported that direct radiation-induced damage and fibrosis may impair lymphatic drainage and antitumor immunity. Early reports have demonstrated a remarkable pathological complete response (pCR) rate of 77.8% with lymph node-sparing short-course radiotherapy (25 Gy in 5 fractions) in locally advanced rectal cancer. In metastatic colorectal cancer, single-fraction high-dose irradiation (6-8 Gy) has been shown to induce robust abscopal effects. Based on these findings, our study aims to evaluate whether lymph node-sparing hypofractionated radiotherapy (25 Gy/5F or 24 Gy/4F) followed sequentially by chemotherapy and PD-1 blockade can increase the pCR rate, improve tolerability, and ultimately enhance outcomes in patients with pMMR/MSS high-risk locally advanced colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signs a written informed consent form.
2. Age ≥ 18 and ≤ 75 years at enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy > 2 years.
5. Histologically confirmed colon adenocarcinoma (without squamous or sarcomatoid components).
6. Tumor biopsy by immunohistochemistry indicating pMMR, i.e., MLH1, MSH2, MSH6, and PMS2 all positive, or genomic testing indicating MSS.
7. Per AJCC 8th edition, imaging (contrast-enhanced CT or contrast-enhanced MRI) shows T4 and/or N+ disease (stage IIB-III).
8. Prior to enrollment, the subject must be evaluated by a surgery attending physician responsible for the operation, based on medical history, to confirm eligibility for R0 resection with curative intent.
9. No prior systemic or local antitumor therapy for rectal cancer before study treatment, including radiotherapy, chemotherapy, immunotherapy, biologics, or small-molecule targeted therapy.
10. Subject agrees to collection and study use of required tumor tissue and peripheral blood specimens during screening and throughout the study.
11. Adequate organ function:

    a) Hematologic (no blood components or hematopoietic growth factors within 7 days before starting study treatment): i. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L (1,500/mm³); ii. Platelets ≥ 100 × 10⁹/L (100,000/mm³); iii. Hemoglobin ≥ 90 g/L. b) Renal: i. Calculated creatinine clearance (CrCl) ≥ 50 mL/min using the Cockcroft-Gault formula: CrCl (mL/min) = {(140 - age) × weight (kg) × 0.85} / [72 × serum creatinine (mg/dL)] ii. Urine protein < 2+ or 24-hour urine protein < 1.0 g. c) Hepatic: i. Total bilirubin (TBil) ≤ 1.5 × ULN; ii. AST and ALT ≤ 2.5 × ULN; iii. Serum albumin (ALB) ≥ 28 g/L. d) Coagulation: i. INR and aPTT ≤ 1.5 × ULN. e) Cardiac: i. Left ventricular ejection fraction (LVEF) ≥ 50%.
12. Women of childbearing potential (WOCBP) must have a urine or serum pregnancy test within 3 days prior to starting study treatment (if the urine test cannot be definitively interpreted as negative, a serum test is required; the serum result prevails) and the result must be negative. If a WOCBP has sexual intercourse with a non-sterilized male partner, she must begin using an acceptable contraceptive method from screening and agree to continue contraception for 120 days after the last dose of study drug; whether contraception can be discontinued thereafter should be discussed with the investigator. Periodic abstinence and calendar/rhythm methods are unacceptable.

    1. WOCBP are defined as females who have not undergone surgical sterilization (i.e., bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy) and have not been postmenopausal (amenorrhea for ≥12 consecutive months without an alternative medical cause, with serum FSH in the postmenopausal range).
    2. A highly effective method of contraception is one with a low failure rate when used consistently and correctly (e.g., <1% per year). Not all methods are highly effective. Barrier methods alone are not acceptable; WOCBP must at minimum use a hormonal contraceptive (e.g., oral contraceptives) to ensure no pregnancy occurs.
13. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study requirements.

    ------

Exclusion Criteria:

1. Suspicious metastatic lesions or the presence of unresectable locally advanced disease, regardless of stage.
2. Malignancy other than colorectal cancer within 5 years prior to enrollment. Subjects cured by local therapy for other malignancies (e.g., basal or squamous cell skin cancer, superficial bladder cancer, ductal carcinoma in situ) are not excluded.
3. Receipt of any investigational drug or device within 4 weeks prior to the first dose of study drug.
4. Intestinal obstruction, perforation, gastrointestinal bleeding, or other conditions requiring emergency surgery.
5. Multiple primary colorectal cancers.
6. Prior radiotherapy to the pelvis or abdomen.
7. Inability to swallow tablets, malabsorption syndrome, or any condition that affects gastrointestinal absorption.
8. Any prior systemic or local antitumor therapy for locally advanced colon cancer, including curative surgery, chemotherapy, radiotherapy, immunotherapy (including immune checkpoint inhibitors/agonists or cellular immunotherapy), biologics, or small-molecule targeted therapy.
9. Nonspecific immunomodulatory therapy within 2 weeks before study treatment (e.g., interleukins, interferons, thymosin, tumor necrosis factor; excluding IL-11 used for thrombocytopenia); antitumor-indicated traditional Chinese herbal medicines or patent medicines within 1 week before study treatment.
10. Active autoimmune disease requiring systemic therapy within the past 2 years (e.g., with disease-modifying agents, corticosteroids, or immunosuppressants). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) is not considered systemic therapy.
11. History of or current non-infectious pneumonitis requiring systemic corticosteroids, or a history of interstitial lung disease.
12. History of significant bleeding tendency or coagulopathy; prior or current long-term anticoagulation (e.g., atrial fibrillation with CHADS₂ score ≥ 2).
13. Uncontrolled comorbid conditions, including but not limited to decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, or psychiatric/social conditions that would limit compliance with study requirements or ability to provide written informed consent.
14. History of myocarditis, cardiomyopathy, or malignant arrhythmias. Within 12 months prior to study treatment: unstable angina requiring hospitalization, congestive heart failure, or vascular disease (e.g., aortic aneurysm requiring surgical repair or peripheral venous thrombosis), or other cardiac damage that may affect evaluation of study-drug safety (e.g., poorly controlled arrhythmias, myocardial infarction or ischemia); within 6 months prior: esophagogastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, enteric fistula, intestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding; within 6 months prior: any arterial thromboembolic event, NCI CTCAE v5.0 grade ≥3 venous thromboembolism, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy; within 1 month prior: acute exacerbation of COPD; current hypertension with SBP ≥160 mmHg or DBP ≥100 mmHg despite oral antihypertensive therapy.
15. Active or past history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) or chronic diarrhea.
16. Serious infection within 4 weeks before study treatment, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective therapy within 10 days before study treatment (excluding antiviral therapy for hepatitis B or C).
17. Major surgery or severe trauma within 30 days before study treatment; minor local surgery within 3 days before study treatment (excluding peripherally inserted central catheter placement).
18. History of immunodeficiency; positive HIV antibody; or current long-term systemic corticosteroid or other immunosuppressive therapy.
19. Known active tuberculosis (TB). Subjects with suspected active TB must be clinically ruled out (e.g., sputum for mycobacteria, chest imaging). Known active syphilis infection.
20. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
21. Untreated active hepatitis B (HBsAg-positive with HBV-DNA > 1,000 copies/mL \[200 IU/mL] or above the assay lower limit). Subjects with hepatitis B must receive antiviral therapy during the study; active hepatitis C (HCV-antibody positive with HCV-RNA above the assay lower limit).
22. Live vaccine within 30 days before study treatment or planned receipt of a live vaccine during the study.
23. Known allergy to any component of the study drugs; history of severe hypersensitivity to other monoclonal antibodies.
24. Known psychiatric illness, substance abuse, alcoholism, or drug dependence.
25. Pregnant or breastfeeding women.
26. Any prior or current disease, therapy, or laboratory abnormality that may confound study results, interfere with full participation, or not be in the subject's best interest to participate.
27. Local or systemic disease not due to malignancy, or tumor-related conditions/symptoms that may confer high medical risk and/or uncertainty in survival assessment, such as leukemoid reaction due to tumor (WBC > 20 × 10⁹/L), cachexia (e.g., >10% body-weight loss within 3 months before screening), or BMI ≤ 18 (BMI = weight[kg] / height [m²]).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2030-08-29 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response(pCR) Rate | From enrollment to 2-4 weeks after surgery
  Evaluate 25Gy/5F or 24Gy/4F node-sparing modified short-course radiotherapy followed by sequential chemotherapy and PD-1 inhibitor as total neoadjuvant therapy can better improve the pathological complete response(pCR) rate in colon cancer.

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | From enrollment to 2-4 weeks after surgery
Tumor downstaging rate | From enrollment to 2-4 weeks after finishing preoperative treatment
R0 resection rate | From enrollment to 2-4 weeks of surgery
3-year overall survival (OS) rate | From enrollment to 3 years after finishing Surgery
Event-Free Survival (EFS) | From enrollment to 3 years after finishing Surgery
3-year distant metastasis rate | From enrollment to 3 years after finishing Surgery
3-year local recurrence rate | From enrollment to 3 years after finishing Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No